CLINICAL TRIAL: NCT01949727
Title: COPD Hospitalization:Examining Pulmonary and Cardiovascular Outcomes in Chronic Obstructive Pulmonary Disease Inpatients (AIM 1). COPD Rehabilitation:Examining the Impact of Early Pulmonary Rehabilitation on Discharged COPD Patients (AIM 2)
Brief Title: Examining Vascular Outcomes in COPD Inpatients (AIM 1) Examining Early Rehabilitation on Discharged COPD Patients (AIM 2)
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Principal Investigator, Michael Stickland, Assistant Professor, University of Alberta
Other Study IDs: Pro00038838; AIHS-CRIO Project Grant (Other: Alberta Innovated Health Solutions (AIHS))
Record Dates: First submitted 2013-09-20; First posted 2013-09-24 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: AECOPD; COPD; Emphysema; Chronic bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AIM 1/AIM 2: AECOPD Admitted Patients: AIM 1:All patients admitted to the hospital (either to Pulmonary or General Medicine) will be recruited to enroll in this observational study. No specific intervention is planned for this group.
  AIM 2: All patients admitted to the pulmonary ward for an AECOPD, including those who have completed Aim 1, will be offered participation into this arm of the study. Pulmonary rehabilitation will be conducted through the Breathe Easy Program at the Centre for Lung Health.
  Interventions: Other: AIM 2: Pulmonary Rehabilitation

INTERVENTIONS:
Other: AIM 2: Pulmonary Rehabilitation — Patients exercise 2 hours per session which includes aerobic exercise (20-40 minutes per session) as well as strength training. All exercise is carefully tracked by trained Respiratory or Physical Therapists. Patients also receive education from a multi-disciplinary team aimed at patient self-management.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a chronic lung disease primarily caused by smoking. COPD creates a tremendous burden to the healthcare system, as disease exacerbations result in frequent, prolonged hospitalizations. While originally considered a disease specific to the lung, data have shown that COPD is associated with substantial cardiovascular (CV) morbidity and mortality. Exacerbations of COPD requiring hospitalization result in marked patient deterioration, and heightened CV risk. The cause of the increased CV risk with stable COPD, and the exaggerated CV risk during exacerbations of the disease are unknown; however, it may be due to chronic inflammation which is exacerbated with a flare-up of the disease, and/or chronic inactivity which is similarly worsened with bed-rest during a hospitalization. Despite the impact of COPD on healthcare, there are relatively few studies examining how COPD inpatient care impacts on patient outcomes, inflammation and CV risk. Disease management programs, such as pulmonary rehabilitation and patient self-management education, are part of guideline therapy for COPD; however, these are not regularly implemented following a hospitalization, and how these interventions affect patient outcomes, behavior, physical activity, inflammation and CV risk have not been well studied. The proposed long-term project will examine how typical inpatient COPD care, and how early referral to chronic disease management programs after hospital discharge, affect patient outcomes. This grant brings together an outstanding group of researchers who have the necessary clinical, content and methodological expertise to successfully complete this work. These studies will provide invaluable information about inpatient and outpatient management for a disease which has a tremendous impact on healthcare.

DETAILED DESCRIPTION:
AIM 1:

Purpose: To examine pulmonary and cardiovascular outcomes in COPD patients from the time of their acute hospital admission until discharge.

Rationale: AECOPD is associated with systemic inflammation, prolonged bed-rest and increased CV risk. Proper medical management strategies such as appropriate systemic corticosteroids, mobilization, and bedside education may reduce systemic inflammation and improve vascular function, while improving patient self-efficacy and health outcomes and reducing hospital length of stay (LOS).

Hypothesis: Treatment-specific factors such as pharmacological management, patient education and inpatient mobilization will affect LOS, as well as pulmonary and cardiovascular outcomes at discharge.

Study Design: For this cross-sectional study, consecutive patients admitted to the University of Alberta Hospital Pulmonary ward with a diagnosis of an AECOPD (with BNP <500 pg/ml and Troponin <1.0 mcg/L), not requiring ventilatory support in the form of non-invasive ventilation (NIV), will be approached for recruitment. In-hospital patient management will be left to the discretion of the admitting physician, and will follow the new AHS admission order sets for AECOPD, which are based on current guidelines1. Dr Bhutani assisted in the development of these order sets. The order sets standardize pharmacological and non-pharmacological management of AECOPD; however, variance in patients need and time to delivery of these interventions will be present. Treatment will not be otherwise altered during this study, except the timing of the administration of short acting bronchodilators as it relates to the measurement of arterial stiffness and vascular function. 24 hours after recruitment, the research team will begin collecting patient/clinical treatment information on a daily basis (see Appendix B for list). 48 hours after admission, patients will be given an activity monitor to quantify daily physical activity. On the same day, vascular assessment through the measurement of pulse wave velocity, vascular function, lung function as well as serum markers of systemic inflammation (TNF-alpha, MMP-2, IL-6 and CRP) and exhaled nitric oxide (eNO), will be collected (this is in addition to usual blood work required for patient management). This will be repeated on days 5, 10, day of discharge and day 14 post discharge. Self efficacy and a 6-minute walk test will be performed on the day of discharge and on day 14 following discharge, while three-day physical activity will be determined at 14 days post discharge. BODE index will be determined at discharge and at 14 days post discharge (see Appendix C for data collection schedule).

Subject Selection & Recruitment: All Aims will be registered at (www.clinicaltrials.gov), submitted for approval through the University of Alberta Health Research Ethics Board (HREB), and informed consent will be obtained from each study patient.

Since most of patients with COPD who are hospitalized initially present to, and are assessed in the Emergency Department (ED), they will be recruited from this setting by the ED study team. All patients with a diagnosis of AECOPD who are admitted to the pulmonary ward, meeting the above criteria, will be screened for enrollment. If entered into the study, baseline information (Appendix A) will be collected at that time. Through collaborative and primary ED research activity, Dr Rowe's Emergency Medicine Research Group maintains research nurse coverage for the U of A hospital ED from 07:00 - 23:00 Monday - Friday and 10:00 - 20:00 Saturday and Sunday. These research nurses act as the main recruitment source within the University of Alberta Hospital ED and this site has been a leading Canadian recruitment centre in a number of clinical research studies. Eligible patients with AECOPD will be approached to enter the study as required and informed written consent will be obtained. A Refused, Missed or Otherwise (RMO) excluded database will be maintained to determine the feasibility of a larger study and to assess the generalizability of the enrolled sample to all cases. In the event that a patient presents after research staff hours, the patient will be approached by the research staff to discuss the study and obtain consent and begin collection of all data. AHS data indicates that ~450 COPD patients are admitted at the U of A hospital each year. Dr Rowe's research team has demonstrated success at recruiting through the ED120,121, and therefore recruiting 100 patients over 2 years is feasible

Data Handling: Upon enrollment a data collection form (Appendix A) will be completed for all patients by the ED research team. The research team will collect patient/clinical treatment information daily (see Appendix B), and outcome data per protocol (see Appendix C).

Data Analysis: All data will be entered into a custom-developed secure anonymized database. Data analyses will be performed using StataCorp. 2009. Stata Statistical Software: Release 11 (College Station, TX: StataCorp LP). Continuous data will be reported as means and standard deviations (SD) or median and interquartile ranges (IQR). Chi-square testing will be used for bi-variable analyses of dichotomous variables; continuous variables will be compared using t-tests or Mann-Whitney tests. Two-tailed results p < 0.05 will be considered statistically significant. The influence of patient characteristics and treatment factors on the dependent variables (i.e. inflammation, vascular function, self efficacy and LOS) will analyzed through a multiple linear or logistic regression models as appropriate. For the linear regression model, clinically relevant and statistically significant (at the p < 0.1 level) independent variables will be included. For the logistic regression model, several dependent variables will be explored; clinically relevant and statistically significant (at the p < 0.1 level) independent variables will be included.

Sample size: A convenience sample of COPD patients will be recruited and efforts will be made to provide reasonable confidence intervals on important variables and outcomes; a minimum sample size of 100 COPD cases will be collected. This will be sufficient for multiple regression analyses including up to 10 predictors and would provide narrow 95% confidence intervals (CI) for variable estimates of ~10% for mid-range variables and 6%. for extreme-range variables.

AIM 2:

Purpose: To examine the impact of early PR following hospital discharge on QoL, pulmonary/CV outcomes and AECOPD hospitalizations.

Rationale: In addition to typical improvements in QoL and exercise tolerance, studies have shown that PR increases self-efficacy, physical activity while reducing CV risk in stable COPD patients. Patients recently discharge from hospital following AECOPD represent the sickest patients with greatly reduced QoL, exercise tolerance, self-efficacy and physical activity and greatly elevated CV risk. Exactly how these improve with PR reduce CV risk and hospitalizations following PR requires examination.

Hypothesis: Patients who receive early PR will have improved QoL, pulmonary/CV outcomes and less hospitalizations for COPD in the 6 months following hospital discharge. PR will improve self efficacy, physical activity and QoL while reducing CV risk as compared to usual care.

Study Design & Subject Recruitment: All patients admitted to the pulmonary ward for an AECOPD, including those who have completed Aim 1, will be offered participation into this arm of the study. Patients found to have an acute cardiac injury during admission, mobility issues or residence outside the greater Edmonton area will be excluded. Consenting patients will be subsequently randomized into one of two groups: early PR versus usual care. Patients randomized to early PR will be enrolled within 1 month of discharge into a PR program, while usual care patients will be followed-up by their most responsible physician as determined by the admitting team. The PR group will be enrolled in the Breathe Easy Program at the Center for Lung Health, and will proceed through the program in a typical fashion. All patients will be followed up 6 months after discharge and will be interviewed to assess disease status, management review and if there has been a history of recurrence or relapse of the AECOPD. Hospital admissions and length of stay data will be obtained through electronic medical records. Patient assessments will include: quality of life, 6min walk, dyspnea, self-efficacy, physical activity, pulse wave velocity, vascular function, systemic inflammation (TNFα, MMP-2, IL-6 and CRP) and FeNO. All data will be collected before, immediately after and 6month after PR. The control group will have the same data collected at the same scheduled time. See above for descriptions of methods.

Data Handling: Data will be entered onto a secure anonymized database.

Data Analysis: The influence of PR on QoL, 6min walk, dyspnea, self-efficacy, physical activity, pulse wave velocity, vascular function, systemic inflammation and eNO will be analyzed using a multivariate mixed-model MANOVA with treatment (PR vs. usual care) being a fixed between-group variable and time (pre, immediate post, 6months post) as a repeated variable.

Sample size: Based on previous work84,95,96,101-105, a sample size of 50 in each group (100 total) will be sufficient to detect a between-group differences in QoL, 6min walk, PWV, dyspnea and hospital readmission rates following PR (α=0.05, β=0.8). Based on our recent work, this sample could detect a 10% difference in physical activity following PR (α=0.05, β=0.8). One hundred patients will also to allow for stratification of physiological and psychological responses with PR.

ELIGIBILITY:
AIM 1:

Inclusion Criteria - Diagnosis of AECOPD who are admitted to the pulmonary ward at the University of Alberta Hospital

Exclusion Criteria

* Age >85
* Cancer Diagnosis/Treatment
* End Stage/Palliative Care
* Dementia
* Hypoxia or respiratory failure impacting ability to consent
* Troponin >1.0
* BNP > 500
* AECOPD not primary diagnosis
* Not admitted to hospital
* Language barrier
* Barriers to follow up

NOTE: Patients with dementia and difficulty with communicating in English are excluded because the questionnaires used have only been validated in English-speaking coherent patients.

AIM 2:

Inclusion Criteria

- Diagnosis of AECOPD who are admitted to the pulmonary ward at the University of Alberta Hospital

Exclusion Criteria

* Age >85
* Cancer Diagnosis/Treatment
* End Stage/Palliative Care
* Dementia
* Hypoxia or respiratory failure impacting ability to consent
* Troponin >1.0
* BNP > 500
* AECOPD not primary diagnosis
* Not admitted to hospital
* Language barrier
* Barriers to follow up
* Mobility issues impacting ability to participate in pulmonary rehabilitation

NOTE: Patients with dementia and difficulty with communicating in English are excluded because the questionnaires used have only been validated in English-speaking coherent patients.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes all English-speaking patients who are admitted to a Pulmonary ward with a diagnosis of Acute Exacerbation of COPD after presenting to ED.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Change in Inflammatory markers | within 24 hours of Admission, within 24 hours of hospital discharge, 14 day follow up
  CRP: C-reactive protein is a non-specific serum marker of inflammation (range <8 is normal)
Change in Vascular Function | Within 24 hours of Admission, within 24 hours of hospital discharge, 14 day follow up
  Vascular Function assessed using EndoPat; RHI: Reactive Hyperemia Index
Change in Arterial Stiffness | Within 24 hours of Admission, within 24 hours of hospital discharge, 14 day follow up
  Pulse wave velocity assessed using Complior

SECONDARY OUTCOMES:
Length of Stay (LOS) | up to 30 days
  Length of stay in the hospital to the point where the patient is stable from the COPD perspective. Patients with LTC needs may stay beyond the designated hospitalization due to care needs.
Readmission-All Cause | up to 1 year
  All cause hospital readmission rates
Readmission-AECOPD | up to 1 year
  AECOPD hospital readmission rates
Change in Physical Activity | Within 24 hours of Admission, within 24 hours of hospital discharge, 14 day follow up
  Step count assessed using a triaxial accelerometer
Change in Inflammatory marker (IL-6) | Within 24 hours of Admission, within 24 hours of hospital discharge, 14 day follow up
  IL-6: is an interleukin that acts as both a pro-inflammatory and anti-inflammatory cytokine.
Inflammatory marker (TNF-alpha) | 14 days
  TNF-alpha
Inflammatory Marker (MMP-2) | 14 days
  MMP-2
Quality of Life (QoL) | 14 days
  CAT MMRC SGHRQ
Immunoglobulin Marker (IgG) | Within 24 hours of Admission
  IgG
Immunoglobulin Marker (IgM) | Within 24 hours of Admission
  IgM
Immunoglobulin Marker (IgA) | Within 24 hours of Admission
  IgA

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stickland, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Fuhr DP, Brotto AR, Rowe BH, Bhutani M, Rosychuk RJ, Stickland MK. Examining changes in vascular function, arterial stiffness and systemic inflammation during hospitalization and recovery from an acute exacerbation of chronic obstructive pulmonary disease. Sci Rep. 2023 Jul 28;13(1):12245. doi: 10.1038/s41598-023-39001-z. PMID 37507427